CLINICAL TRIAL: NCT03097094
Title: Precision Allergy: Separate Allergies to Male and Female Dogs
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Copenhagen Studies on Asthma in Childhood (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Diagnostic
Other Study IDs: Dog allergy
Record Dates: First submitted 2017-03-24; First posted 2017-03-31 (Actual); Last update posted 2022-11-15 (Actual); Status verified 2022-11

CONDITIONS: Allergy; Dander
Keywords: Dog allergy; Can f 5; Male dog; Female dog; Allergen components
MeSH Terms: conditions — Hypersensitivity

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Male dog (Active Comparator): Male dog extract used for skin prick test and conjunctival provocation
  Interventions: Diagnostic Test: Male dog
- Female dog (Active Comparator): Female dog extract used for skin prick test and conjunctival provocation
  Interventions: Diagnostic Test: Female dog

INTERVENTIONS:
Diagnostic Test: Male dog — Male dog extract
  Arms: Male dog
Diagnostic Test: Female dog — Female dog extract
  Arms: Female dog

SUMMARY:
A new male-specific dog-allergen-component has been found (Can f 5) which indicates possible differences in allergic reactions to male and female dogs. This has not yet been tested in real life.

The aim is to test if sensitization only to the male-dog specific allergen-component, Can f 5, results in a positive skin prick test (SPT) to male dog extract and not female dog extract. In addition, the investigators want to investigate if allergic symptoms only occur when exposed to the male dog extract by conjunctival provocation.

ELIGIBILITY:
Inclusion Criteria:

* Participants in the COPSAC 2000 cohort
* Positive component test (>0.3 ISU) to Can f 1, Can f 2, Can f 3 or Can f 5

Exclusion Criteria:

* Uncontrolled asthma
* Eye-surgery within the past 6 months
* Antihistamine allergy
* and others

Min Age: 15 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2017-03-24 (Actual); Primary Completion 2017-09-01 (Actual); Study Completion 2019-01-09 (Actual)

PRIMARY OUTCOMES:
Male vs. female dog SPT in Can f 5 mono sensitized patients | 6 months
  In the patients that have a positive SPT (> 2mm) to dog and are monosensitized to the Can f 5 component, the investigatiors want to compare the reaction to SPT (pos/neg) to male vs. female dog extract in the same patient using logistic regression analysis with mixed effects to account for repeated measures.

SECONDARY OUTCOMES:
Male vs. female dog conjunctival provocation in Can f 5 mono sensitized patients | 6 months
  In the patients that have a positive SPT (> 2mm) to dog and are monosensitized to the Can f 5 component, the investigatiors want to compare the reaction to conjunctival provocation (positive/negative) to male vs. female dog extract in the same patient using logistic regression analysis with mixed effects to account for repeated measures.
Male vs. female dog SPT in dog poly sensitized patients | 6 months
  In the patients that have a positive SPT (> 2mm) to dog and are sensitized to the Can f 1, 2 and/or 3 component, the investigatiors want to compare the reaction to SPT (pos/neg) to male vs. female dog extract in the same patient using logistic regression analysis with mixed effects to account for repeated measures.
Male vs. female dog conjunctival provocation in dog poly sensitized patients | 6 months
  In the patients that have a positive SPT (> 2mm) to dog and are sensitized to the Can f 1, 2 and/or 3 component, the investigatiors want to compare the reaction to conjunctival provocation (pos/neg) to male vs. female dog extract in the same patient using logistic regression analysis with mixed effects to account for repeated measures.
Can f 5 vs. SPT size | 6 months
  To investigate the correlation between specific Immunoglobulin E (sIgE) level to the Can f 5 component and the SPT wheal size to the male dog extract using a general linear model.
Can f 5 vs. conjunctival provocation | 6 months
  To investigate the correlation between sIgE level to the Can f 5 component and the threshold of reaction to the male dog extract at the conjunctival provocation, using a general linear model.
SPT vs. conjunctival provocation | 6 months
  To investigate the correlation between SPT wheal size to the male dog extract and the threshold of reaction to the male dog extract at the conjunctival provocation, using a general linear model.

CONTACTS AND LOCATIONS:
Overall Officials: Klaus Bønnelykke, MD, PhD, Principal Investigator — Copenhagen Studies on Asthma in Childhood
Locations (1):
- Copsac, Dbac, Gentofte Municipality, Copenhagen, Denmark

IPD SHARING:
Plan to Share IPD: No